CLINICAL TRIAL: NCT01132443
Title: A Phase 1, Single Center, Randomized, Open-Label Study to Evaluate the Bioavailability of Clindamycin From Clindamycin 1%-Benzoyl Peroxide 3% Gel, Topical Gel (Clindamycin 1%- Benzoyl Peroxide 5%), and Once Daily Gel (Clindamycin 1%-Benzoyl Peroxide 5%) in Subjects With Acne Vulgaris
Brief Title: W0261-101: A Phase 1, Single Center, Randomized, Open-Label Study to Evaluate the Bioavailability of Clindamycin From Clindamycin 1%-Benzoyl Peroxide 3% Gel, Topical Gel (Clindamycin 1%- Benzoyl Peroxide 5%), and Once Daily Gel (Clindamycin 1%-Benzoyl Peroxide 5%) in Subjects With Acne
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 115902
Record Dates: First submitted 2010-05-24; First posted 2010-05-28 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin; Benzoyl Peroxide; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Clindamycin 1%-Benzoyl Peroxide (BPO) 3% Gel, (Experimental): Apply topically once daily; clindamycin (CLN); benzoyl peroxide (BPO); methylparaben-free (MPF)
  Interventions: Drug: Clindamycin 1%-Benzoyl Peroxide (BPO) 3% Gel,
- Duac/ formulation 1 (Active Comparator): Apply topically once daily, Topical Gel (CLN 1%-BPO 5%), methylparaben-preserved
  Interventions: Drug: Clindamycin 1%-Benzoyl Peroxide (BPO) 3% Gel,
- Duac/ formulation 2 (Active Comparator): Apply topically once daily, Duac Once Daily Gel (CLN 1%-BPO 5%), MPF
  Interventions: Drug: Clindamycin 1%-Benzoyl Peroxide (BPO) 3% Gel,

INTERVENTIONS:
Drug: Clindamycin 1%-Benzoyl Peroxide (BPO) 3% Gel, — Apply topically once daily

SUMMARY:
This study was conducted to determine if the bioavailability of clindamycin and its metabolite clindamycin sulfoxide are altered by the concentration of BPO or the absence of methylparaben. This study compared the investigational study product and 2 marketed products:

* CLN 1%-BPO 3% Gel (clindamycin 1%-BPO 3%), methylparaben-free
* Topical Gel (clindamycin 1%-BPO 5%), methylparaben-preserved (Topical Gel-MP)
* Once Daily Gel ((clindamycin 1%-BPO 5%), methylparaben-free (Topical Gel-MPF)

DETAILED DESCRIPTION:
Clindamycin and benzoyl peroxide (BPO) are both well-known treatments for acne vulgaris (acne) and are available as single-entity and fixed-dose combination products. The same excipients are used in the gel vehicle formulations, except inclusion of the preservative methylparaben in the vehicle is dependent on geographic region. While these products have been shown to be well tolerated, effective combination therapies for acne, concentration-dependent cutaneous irritation has been associated with the use of BPO.

Clindamycin 1%-benzoyl peroxide 3% gel (CLN 1%-BPO 3%) for the topical treatment of acne was developed. CLN 1%-BPO 3% contains the same concentration of clindamycin and a lower concentration of BPO than currently-marketed products, and CLN 1%-BPO 3% is formulated without methylparaben.

A study to evaluate the plasma concentrations of clindamycin and its metabolites after topical gel was applied once daily for 4 weeks in subjects with moderate-to-severe acne showed that the absorption of clindamycin and its metabolite clindamycin sulfoxide were comparable between Topical Gel and a representative single entity product with the same clindamycin concentration. An in vitro skin penetration study demonstrated that there were no significant differences in the delivery of clindamycin in and through the skin following application of either CLN 1%-BPO 3% or topical gel; therefore, the presence of BPO in the formulation at either 3% or 5% did not have an effect on the percutaneous absorption of clindamycin.

Benzoyl peroxide has been shown to be absorbed by the skin where it is converted to benzoic acid. Following topical application, less than 2% of the dose enters systemic circulation as benzoic acid. The transepidermal delivery of BPO is dependent on concentration and no systemic toxicity is expected due to rapid renal clearance of benzoic acid. Benzoic acid is frequently utilized as a preservative or to adjust the pH in food, cosmetics, and medicinal products; therefore, the limited systemic absorption from CLN 1%-BPO 3% is not expected to notably increase exposure to benzoic acid. Due to the low potential for systemic toxicity and the limited utility of assessing plasma concentrations of benzoic acid, the systemic exposure was not evaluated in this study.

Systemic exposure to clindamycin has been associated with severe cases of diarrhea, bloody diarrhea and colitis (including pseudomembranous colitis), which could be fatal. Several studies conducted with single-entity and fixed-combination topical clindamycin-containing products have determined that systemic absorption of clindamycin is low; however, there have been documented cases of colitis after topical administration of clindamycin phosphate. Clindamycin phosphate is rapidly hydrolyzed in vivo to clindamycin, the active parent compound. Topical application of Clindagel (clindamycin phosphate 1% gel) equivalent to 3 to 12 grams once daily for 5 days resulted in peak plasma clindamycin concentrations that were less than 5.5ng/mL. Multiple topical applications of Cleocin T (clindamycin phosphate at a concentration equivalent to 10mg/mL) resulted in clindamycin serum levels ranging from 0 to 3 ng/mL. The mean systemic bioavailability of clindamycin is less than 1%.

As there exists a potential for different topical formulations to have greater systemic exposure to the active ingredients than currently marketed products, this study was conducted to determine if the bioavailability of clindamycin and its metabolite clindamycin sulfoxide are altered by the concentration of BPO or the absence of methylparaben. This study compared the investigational study product and 2 marketed products:

* CLN 1%-BPO 3% Gel (clindamycin 1%-BPO 3%), methylparaben-free
* Topical Gel (clindamycin 1%-BPO 5%), methylparaben-preserved (Topical Gel-MP)
* Once Daily Gel ((clindamycin 1%-BPO 5%), methylparaben-free (Topical Gel-MPF)

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding and willing to provide signed and dated written voluntary informed consent (and HIPAA authorization) before any protocol-specific procedures were performed. Subjects under the legal age of consent in the state where the study was conducted must have provided assent and have had the written informed consent of a parent or guardian.
* Male or female 12 to 45 years of age at time of consent.
* Moderate-to-severe facial acne, defined as an ISGA score of 3 or greater.
* Able to complete the study and to comply with study instructions.
* Sexually-active females of childbearing potential participating in the study must have agreed to use a medically-acceptable method of contraception while receiving protocol-assigned product. A woman of childbearing potential was defined as one who is biologically capable of becoming pregnant, including perimenopausal women who are less than 2 years from their last menses. Acceptable contraceptive methods included the following:
* Hormonal contraception, including oral, injectable, or implantable methods started at least 3 months prior to screening. If hormonal contraception was started less than 3 months prior to screening, then a form of nonhormonal contraception should have been added until the third continuous month of hormonal contraception had been completed.
* Two forms of reliable nonhormonal contraception, to include the use of either an intrauterine device plus a reliable barrier method or 2 reliable barrier methods. Reliable barrier methods include condoms or diaphragms. A cervical cap is also a reliable barrier method, provided the female subject has never given birth vaginally. The combined use of a condom and spermicide constitute 2 forms of acceptable nonhormonal contraception, provided that they are both used properly. The use of spermicide alone and the improper use of condoms are inferior methods of contraception. Subjects with surgical sterilization, including tubal sterilization or partner's vasectomy, must have used a form of nonhormonal contraception. A barrier method or sterilization plus spermicide was acceptable.
* Women who were not currently sexually active must have agreed to use a medically-acceptable method of contraception should they have become sexually active while participating in the study.

Exclusion Criteria:

* Female who was pregnant, trying to become pregnant, or breast feeding.
* Participation in any investigational study within 4 weeks of Day 1 or who were scheduled to participate in another investigational study in the next 2 weeks.
* Used prohibited medications within specified time period before Day 1.
* Currently using any medication that, in the opinion of the investigator, may affect the evaluation of the study product or place the subject at undue risk.
* History or evidence of skin conditions other than acne (eg, eczema, rosacea, seborrheic dermatitis, birthmarks, tattoos) that would interfere with study evaluations.
* History or presence of regional enteritis or inflammatory bowel disease (eg, ulcerative colitis, pseudomembranous colitis, chronic diarrhea, celiac disease, Crohn's disease, or history of antibiotic-associated colitis) or similar symptoms.
* Had any major illness within 4 weeks of Day 1.
* Anticipated need for surgery or hospitalization during the study.
* Blood donation, or equivalent blood loss (~480 mL), within 3 months of Day 1.
* Anemia or any other systemic disease condition for which a loss of 120 mL of blood over a 1-week period may put the subject at undue risk.
* Considered immunocompromised.
* Currently suffering from any disease or condition that, in the opinion of the investigator, may affect the evaluation of the study product or place the subject at undue risk.
* Current smoker or smoker with less than 4 weeks abstinence from smoking and nicotine-containing products.
* Anticipated need to engage in activities or exercise that would cause profuse sweating during the study.
* Required or desired excessive or prolonged exposure to ultraviolet light (eg, sunlight, or tanning beds) during the study.
* Clinically relevant history of or current evidence of abuse of alcohol or other drugs.
* History of known or suspected intolerance, hypersensitivity, or allergic reaction to any of the ingredients of the study products, including clindamycin and BPO.
* Considered unable or unlikely to attend the necessary visits.
* Lived in the same household as currently enrolled subjects.
* Employee of the investigator, clinical research organization, or Stiefel who was involved in the study, or an immediate family member (eg, partner, offspring, parents, siblings, or sibling's offspring) of an employee who was involved in the study.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2010-05-06 (Actual); Primary Completion 2010-06-12 (Actual); Study Completion 2010-06-12 (Actual)

PRIMARY OUTCOMES:
Clindamycin plasma concentrations | Baseline to Day 6
  Plasma concentrations of clindamycin in subjects with acne vulgaris

SECONDARY OUTCOMES:
Clindamycin sulfoxide plasma concentrations | Baseline/Day 1, Day 2, 3, 4, and 5 (pre-dose and 1, 2, 4, 6, 8, 12, and 24 hours post dost - Day 6)
  Plasma concentrations of clindamycin sulfoxide in subjects with acne vulgaris

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Jones TM, Jasper S, Alio Saenz AB. Bioavailability of Clindamycin From a New Clindamycin Phosphate 1.2%-Benzoyl Peroxide 3% Combination Gel. Clin Pharmacol Drug Dev. 2013 Jan;2(1):33-47. doi: 10.1002/cpdd.7. Epub 2013 Mar 4. PMID 27121558
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 115902 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115902?search=study&study_ids=115902#rs
- Available data/document: Statistical Analysis Plan: 115902 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115902 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115902 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115902 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115902 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115902 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115902 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register